CLINICAL TRIAL: NCT06785389
Title: Influence of Preoperative Fear on Pain and Postoperative Outcomes
Acronym: POSPoFe
Status: Recruiting | Type: Observational
Sponsor: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Ángel Becerra-Bolaños, MD PhD, Principal Investigator, Dr. Negrin University Hospital
Other Study IDs: 2024-472-1
Record Dates: First submitted 2025-01-16; First posted 2025-01-21 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Fear; Pain Management; Anxiety; Complications of Surgical Procedures or Medical Care
Keywords: preoperative fear; postoperative pain; postoperative outcomes; preoperative anxiety
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients scheduled for surgery: Patients undergoing surgery under general anesthesia with hospital admission.
  Interventions: Diagnostic Test: Fear of anesthesia, surgery and hospitals scale; Diagnostic Test: State-Trait Anxiety Inventory; Diagnostic Test: Nummerical Rating Scale for postoperative pain

INTERVENTIONS:
Diagnostic Test: Fear of anesthesia, surgery and hospitals scale — The day before surgery, patients will be interviewed using the scales of Fear of anesthesia, surgery and hospitals.
Diagnostic Test: State-Trait Anxiety Inventory — The day before surgery, patients will be interviewed using the State-Trait Anxiety Inventory
Diagnostic Test: Nummerical Rating Scale for postoperative pain — In the first postoperative day, patients will be monitored using the Nummerical Rating Scale, which will assess postoperative pain.
  Other Names: Nummerical Rating Scale

SUMMARY:
Fear of anesthesia plays a crucial role in the perioperative setting and can negatively affect recovery. The main objective is to assess the relationship between fear of anesthesia, surgeries, and hospitals and poorer postoperative pain control in patients undergoing scheduled surgery, as well as to relate preoperative anxiety to postoperative analgesic assessment in this population.

This is a prospective observational study including 138 patients scheduled for surgery.

DETAILED DESCRIPTION:
Fear is a response that arises in the face of immediate threats, such as medical procedures, while anxiety is related to uncertainty about treatment and prognosis. These factors can negatively affect recovery. Assessing anxiety levels using specific tools may be essential to predict clinical outcomes and facilitate patient recovery after surgery.

This prospective observational study will assess the relationship between fear of anesthesia, surgeries, and hospitals and poorer postoperative pain control in patients undergoing scheduled surgery. It will also relate preoperative anxiety to postoperative analgesic assessment in this population.

Disease or disorder under study: Fear of anesthesia and postoperative pain control using two preoperative questionnaires. Patients will be followed up until discharge to assess postoperative pain and postoperative outcomes. Considering that the estimated percentage of fear is around 10%, with a 95% confidence interval and a 5% error margin, 138 patients are needed to accurately estimate its prevalence in the population.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years old scheduled for surgery with admission during the study period will be included.
* Verbal and written informed consent.

Exclusion Criteria:

* Minors
* Cognitive impairment
* Patients not being able to understand and respond to preoperative questionnaires
* Patients not being able to respond to postoperative pain assessment
* Patients not giving informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing scheduled surgery with general anesthesia requiring hospital admission during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain using Nummerical Rating Scale | 24 hours
  In the first postoperative day, patients will be monitored using the Nummerical Rating Scale, which will assess postoperative pain, from 0 (no pain) to 10 (maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: Undecided